CLINICAL TRIAL: NCT07133295
Title: Long-Term Efficacy and Safety of Once-Weekly Levothyroxine Regimen in Hypothyroid Patients: A Three-Year Follow-Up Study
Brief Title: Long-Term Efficacy and Safety of Once-Weekly Levothyroxine Regimen in Hypothyroid Patients
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hany Ahmed Mohamed, lecturer of internal medicine department, Sohag University
Other Study IDs: Soh-Med-25-4--7PD
Record Dates: First submitted 2025-05-16; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-04

CONDITIONS: Hypothyroidism
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 patients who will continue to take L-T4 on standard daily basis.
- Group 2 patients who will switch to once weekly dosing

SUMMARY:
Hypothyroidism is a prevalent endocrine disorder characterized by insufficient production of thyroid hormones. Traditional treatment involves daily administration of levothyroxine (L-T4), which can be challenging for some patients due to adherence issues. Recent studies have explored the efficacy of once-weekly L-T4 regimens, suggesting that they may provide a viable alternative for patients struggling with daily dosing The safety profile of once-weekly L-T4 has also been a focus of recent research. Evidence indicates that this regimen is associated with minimal side effects and is well-tolerated by patients. A comparative study found that once-weekly L-T4 did not result in significant adverse effects compared to daily dosing, reinforcing its potential as a safe treatment option

DETAILED DESCRIPTION:
Hypothyroidism is a prevalent endocrine disorder characterized by insufficient production of thyroid hormones. Traditional treatment involves daily administration of levothyroxine (L-T4), which can be challenging for some patients due to adherence issues. Recent studies have explored the efficacy of once-weekly L-T4 regimens, suggesting that they may provide a viable alternative for patients struggling with daily dosing. A study published in 2023 demonstrated that once-weekly L-T4 is effective in maintaining euthyroidism in patients with treatment-refractory hypothyroidism.

The safety profile of once-weekly L-T4 has also been a focus of recent research. Evidence indicates that this regimen is associated with minimal side effects and is well-tolerated by patients.

Adherence to treatment is crucial for the management of hypothyroidism, and once-weekly regimens may enhance patient compliance. Studies have shown that patients are more likely to adhere to a once-weekly regimen compared to daily dosing, which can lead to improved clinical outcomes. This is particularly relevant for patients with non-adherence issues, as highlighted in recent literature.

ELIGIBILITY:
Inclusion Criteria:

* All included hypothyrodism patients will be euthyroid, and stable on the same L-T4 dose before the start of study.

Exclusion Criteria:

-1- patients with thyroid cancer patients requiring suppressive therapy 2-patients with central hypothyroidism 3- pregnancy, coronary heart disease, arrythmia, chronic heart failure 4-patients with liver cirrhosis, renal failure, acute medical, or surgical illness at the time of evaluation to avoid acute and chronic non-thyroidal illness syndromes.

4- Patients taking any medications known to interfere with levothyroxine absorption or metabolism (calcium and iron supplements, antiepileptic agents, antacids, proton pump inhibitors, and H2blockers)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This a prospective randomized conducted over three years will be including hypothyroid patients attending outpatient clinic, Sohag faculty of medicine, Sohag university, Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the maintenance of euthyroidism,defined as normal thyroid function | From baseline (study enrollment) until 36 months after enrollment. first year :assessments will be conducted 2 months after each dose adjustment in subsequent years assessment conducted quarterly up to end of the study
  Normal thyroid function, assessed via:
  TSH: Normal range [specify, e.g., 0.4-4.0 µIU/mL]
  Free T4: Normal range [specify, e.g., 0.8-1.8 ng/dL]

SECONDARY OUTCOMES:
. Secondary outcomes will include:-1- the incidence of adverse effects(clinical parameters) | 1-Baseline (Day 1) until 24 months 2-Week 8 (2 months post-initial dose adjustment) 3-Every 12 weeks (±7 days) thereafter until study completion (up to 24 months)
  1-Incidence of Adverse Effects:* Clinical parameters:
  1. Heart rate (beats per minute)
  2. Blood pressure (mmHg)
secondary outcome 2-Incidence of Adverse Effects - Laboratory Parameters (Complete Blood Count) | From Baseline (Day 1) until study completion (up to 24 months), assessed at Week 8 (2 months post-initial dose adjustment) and every 12 weeks (±7 days) thereafter.
  Incidence of clinically significant abnormalities in Complete Blood Count Unit of Measure: (e.g., cell counts in cells/µL, hemoglobin in g/dL, hematocrit in %)
secondary outcome. 3- Incidence of Adverse Effects - Laboratory Parameters (Liver Function Tests) | From Baseline (Day 1) until study completion (up to 24 months), assessed at Week 8 (2 months post-initial dose adjustment) and every 12 weeks (±7 days) thereafter.
  Incidence of clinical abnormalities Liver Function Tests(e.g., ALT, AST) U/L
  Unit of Measure: U/L
4-Incidence of Adverse Effects - Laboratory Parameters (Kidney Function Tests) | From Baseline (Day 1) until study completion (up to 24 months), assessed at Week 8 (2 months post-initial dose adjustment) and every 12 weeks (±7 days) thereafter.
  Incidence of clinical abnormalities in Kidney Function Tests (e.g., serum creatinine)
  Unit of Measure: mg/dL
secondary outcome include :-2-Patient Adherence Rates | 1-from baseline(day 1) until 36 months 2-Monthly from Baseline to Week 52 3-- 12 weeks from Week 52 to study completion
  2-Patient Adherence Rates :Measured via self-report, pill counts, or pharmacy refill records. Criteria for adherence (e.g., ≥80% of doses taken).
secondary outcome include:-3. Quality of Life (QoL) Assessments using ThyPRO | 1-From Baseline(day 1) until 36 months after enrollment assessed at Baseline, Week 8, Week 24, Week 52, and every 24 weeks thereafter.
  Thyroid-specific QoL measured using validated questionnaires:
  ThyPRO (Thyroid Patient-Reported Outcome)
  Unit of Measure:
  ThyPRO: Scale scores (0-100)
Quality of Life (QoL) Assessments - SF-36 | From Baseline (day 1)until 36 months Aassessed at Baseline, Week 8, Week 24, Week 52, and every 24 weeks thereafter.
  chang in general quality of life using SF-36 (Short Form Health Survey) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: sara Kasem Abdelal, lecturer, Study Chair — sohag university .faculty of medicine
Locations (1):
- sohag faculty of medicine, Sohag, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided